CLINICAL TRIAL: NCT01366989
Title: INBONE Total Ankle Arthroplasty(TAA)Using Calcaneal Stem Fixation
Status: Terminated | Type: Observational
Why Stopped: The retrospective data review did not provide adequate information to continue the investigation.
Sponsor: Stryker Trauma and Extremities (Industry)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: 08-SJA-001
Record Dates: First submitted 2011-06-02; First posted 2011-06-06 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Arthrodesis; Degenerative Arthritis; Rheumatoid Arthritis; Complications; Arthroplasty, Mechanical
Keywords: Total Ankle Arthroplasty
MeSH Terms: conditions — Ankylosis; Osteoarthritis; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Total Ankle Arthroplasty with calcaneal stem: Patients received the TAA with calcaneal stem between 12/6/05 & 11/13/07 at approximately 28 sites.
  Interventions: Device: Radiographic evaluation of previously implanted patients

INTERVENTIONS:
Device: Radiographic evaluation of previously implanted patients — Radiographs of the ankle
  Other Names: Radiographs of previously implanted patients

SUMMARY:
The primary objective of this study is to evaluate the radiographic outcomes of Total Ankle Arthroplasty in patients having a calcaneal stem.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the radiographic outcomes of patients who have received TAA with the calcaneal stem. Due to the fixation of the stem in the calcaneus, talar component position, osteolysis and bone quality are of interest to the FDA. Specifically, subsidence and/or migration of the talar component, osteolysis as a measure of wear, and bone quality of the talus, cuboid and navicular are to be evaluated in this study. Therefore, the radiographic outcomes of this study aim to assess these parameters

ELIGIBILITY:
Inclusion Criteria:

Patients who will be recruited for participation in this study received the TAA with calcaneal stem between December 6, 2005 and November 13, 2007 at approximately 28 sites.

Exclusion Criteria:

Patients who will be recruited for participation in this study received the TAA with calcaneal stem between December 6, 2005 and November 13, 2007 at approximately 28 sites.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will be recruited for participation in this study received the TAA with calcaneal stem between December 6, 2005 and November 13, 2007 at approximately 28 sites.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2013-06-04 (Actual); Study Completion 2013-06-04 (Actual)

PRIMARY OUTCOMES:
Radiographic Evaluation | Post operarative 1.2 -3.1 years
  Bone quality of the talus, navicular, and cuboid will be assessed on both the lateral and mortise views of the latest follow-up radiographs

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bolognesi, MD, Principal Investigator — Duke University
Locations (1):
- Michael Bolognesi, MD, Durham, North Carolina, United States